CLINICAL TRIAL: NCT03496220
Title: Measuring the Effect of Angulus on Patient-elevation Compliance
Brief Title: Effect of Angulus on Patient-elevation Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angulus, LLC (Industry)
Collaborators: Albert Einstein College of Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 001; 1R43HL131177-01A1 (NIH)
Record Dates: First submitted 2018-04-02; First posted 2018-04-12 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Ventilator Adverse Event; Ventilator Associated Pneumonia; Hospital Acquired Condition; Hospital-acquired Pneumonia; Recumbency; Head-of-bed
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Iatrogenic Disease; Healthcare-Associated Pneumonia

STUDY DESIGN:
Intervention Model Description: Clustered randomized cross over trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Feedback (Experimental): The ICU with feedback will be equipped with display device corresponding to each Angulus device with an interactive software interface which displays the patient's elevation.
  Interventions: Device: Angulus
- No Feedback (Other): The Angulus device will be on the patient but will NOT have the corresponding display data on patient elevation available to nurses.
  Interventions: Device: Angulus

INTERVENTIONS:
Device: Angulus — Feedback on patient recumbency

SUMMARY:
Ventilator-associated events (VAE) are a scourge of critical care settings and hospital systems at large. There is extensive evidence that ventilator-associated pneumonia (VAP) and related VAEs increase mortality rates in critically ill patients by up to 50%, while simultaneously increasing cost of care. C

Best-practice guidelines state that positioning ventilated patients at an angle between 30-45 degrees significantly reduces the potential for VAP and other VAE to develop. While the intent of the guidelines is to govern patient elevation angle, the lack of a mechanism to accurately measure patient elevation requires that nurses rely on the head-of-bed (HOB) protractor - a tool which reflects the angle of the bed, not the patient - to measure compliance. Depending upon the position and posture of the patient in the bed, a patient's elevation angle may be significantly different from the HOB angle. Critical care teams currently rely on built-in HOB protractors and digital inclinometers that measure the angle of the bed not the patient.

Angulus, LLC has developed a dual-component Angulus sensor to fill this gap in critical care technology. Angulus enables critical care practitioners to instantaneously understand a patient's elevation, identify when the patient is outside of the desired 30-45 degree recumbency scope, and efficiently correct the patient's orientation with immediate feedback. Angulus supports real-time minute-to-minute data display as well as longitudinal aggregation of data.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation with any modality (e.g., endotracheal tube, tracheostomy)
* Age between 18 and 75 years

Exclusion Criteria:

* Patients with a known allergy to the encasing materials
* Patients who are advised to be positioned outside of the 30-45 degree scope.
* Patients with any major chest wall abnormalities, or defects, including but not limited to:

  * post-cardiac surgical patients
  * pectus excavatum (or any congenital chest wall deformity)
  * complicated skin and soft tissue infections on the chest wall
  * heart-lung machine systems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Gong, MD, Principal Investigator — Einstein College of Medicine, Division of Critical Care
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ICU A Feedback First, Then no Feedback, and Feedback Last; ICU B No Feedback First, Then Feedback, and No Feedback Last; ICU C: Feedback First, Then No Feedback, and Feedback Last: During the feedback period ICU will be equipped with display device corresponding to each Angulus device with an interactive software interface which displays the patient's elevation.
  In the No Feedback period the Angulus device will be on the patient but will NOT have the corresponding display data on patient elevation available to nurses.
  Angulus: Feedback on patient recumbency
Period: First Intervention
Arm/Group | ICU A Feedback First, Then no Feedback, and Feedback Last | ICU B No Feedback First, Then Feedback, and No Feedback Last | ICU C: Feedback First, Then No Feedback, and Feedback Last
Started | 15 | 4 | 10
Completed | 15 | 4 | 10
Not Completed | 0 | 0 | 0
Period: Second Intervention
Arm/Group | ICU A Feedback First, Then no Feedback, and Feedback Last | ICU B No Feedback First, Then Feedback, and No Feedback Last | ICU C: Feedback First, Then No Feedback, and Feedback Last
Started | 17 | 9 | 11
Completed | 17 | 9 | 11
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | ICU A Feedback First, Then no Feedback, and Feedback Last | ICU B No Feedback First, Then Feedback, and No Feedback Last | ICU C: Feedback First, Then No Feedback, and Feedback Last
Started | 11 | 8 | 5
Completed | 11 | 8 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Feedback | No Feedback | Total
Number analyzed (Participants) | 49 | 41 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 31 | 63
  >=65 years | 17 | 10 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (12.7) | 58.7 (10.1) | 57.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 33 | 22 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 14 | 32
  Not Hispanic or Latino | 31 | 27 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 14 | 31
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 16 | 35
Region of Enrollment [Number; unit: participants]
  United States | 49 | 41 | 90

OUTCOME MEASURES:

1. Primary Outcome: Compliance to Head of Bed Elevation to 30 Degree or More.
Description: Measured as a continuous variable between 0% and 100% compliance.
Time Frame: 3 months
Population: Time spent in evidence based recumbency range comparison.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Feedback | No Feedback
Number analyzed (Participants) | 49 | 41
percentage of time | 37.3 (26.2) | 32.4 (29.3)

ADVERSE EVENTS:
Time Frame: 3 months
Description: No adverse events were noted as a result of participation in the study.
Arm/Group | Feedback | No Feedback
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/41
Other Adverse Events (participants affected / at risk) | 0/49 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT03496220/Prot_SAP_001.pdf